CLINICAL TRIAL: NCT06231485
Title: A Randomized Intervention Trial to Increase Access to Reproductive Health Services Among Adolescents and Young Adults With Intellectual and Developmental Disabilities
Brief Title: Socialization To Enrich Participation & Support Sexuality for Young People With I/DD
Acronym: STEPS2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: City University of New York, School of Public Health (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Institutes of Health INCLUDE Project (Unknown); National Institutes of Health Office of Disease Prevention (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2022-0617; 1R01HD111044-01 (NIH)
Record Dates: First submitted 2023-09-20; First posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Knowledge; Behavior
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Intervention Model Description: Half of the participants will be randomized to receive the socialization and sex education curriculum (STEPS2), and half to the nutrition and physical exercise curriculum (STYH)
Who Masked: Outcomes Assessor
Masking Description: Interviewers (outcomes assessors) are masked to the intervention arm to reduce the potential for bias during the interview process, as all surveys are interviewer-administered.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Socialization and sex education (STEPS2) (Experimental): Weekly virtual one hour one-on-one sessions with Study Health Educator on the STEPS2 curriculum for 6-weeks. Topics include: the human body, decision-making, sexually transmitted diseases, pregnancy, birth control, pregnancy and parenting, and going to the doctor.
  Interventions: Behavioral: STEPS2
- Nutrition and physical activity (STYH) (Other): The comparison curriculum has been shown in a previous study to improve knowledge around nutrition and exercise, but should not change sexual and reproductive health outcomes.
  Weekly virtual one hour group sessions (6-10 participants) with Study Health Educator on the Steps To Your Health (STYH) curriculum for 6-weeks. Topics include: nutrition, exercise, stress management, changing your way of thinking, and behaviors to stay healthy.
  Interventions: Behavioral: STYH

INTERVENTIONS:
Behavioral: STEPS2 — One of the two health education curricula as described in arm/group descriptions.
  Arms: Socialization and sex education (STEPS2)
Behavioral: STYH — One of the two health education curricula as described in arm/group descriptions.
  Arms: Nutrition and physical activity (STYH)

SUMMARY:
The goal of this clinical trial is to test the effectiveness of a 6-week socialization and sex education curriculum (STEPS2) in young people (aged 16-27 years) with intellectual and developmental disabilities (I/DD), including people with Down syndrome.

The main question it aims to answer is:

Does the STEPS2 health education curriculum increase the proportion of individuals who:

1. have had a discussion with a medical professional about their sexual health (including sexually transmitted infection testing for those who are sexually active);
2. know whether they have had the HPV vaccination;
3. have had the HPV vaccination;
4. know what sex is; and
5. know how people get pregnant.

These are the primary outcomes which are being measured one year after study enrollment. Secondary outcomes include knowledge around sexual health and behaviors around contraception and STI prevention among those sexually active at baseline, as well as satisfaction with the intervention.

Participants are randomized to receive either the socialization and sex education curriculum in the experimental group, called the STEPS2 curriculum, or a nutrition and physical exercise curriculum in the comparison group, called Steps To Your Health (STYH).

Participants in the STEPS2 experimental group meet with a health educator in one-on-one individually tailored sessions virtually once a week for one hour for 6 weeks. Participants in the STYH comparison group meet with a health educator in small group sessions of 6-10 participants virtually once a week for one hour for 6 weeks.

Researchers will compare sexual and reproductive health knowledge and behaviors one year after study enrollment to see if the STEPS2 curriculum is effective at increasing knowledge and healthy behaviors.

DETAILED DESCRIPTION:
The goal of this clinical trial is to test the effectiveness of a 6-week socialization and sex education curriculum (STEPS2) among 856 adolescent and young adults (aged 16-27 years) with mild to moderate intellectual or developmental disabilities (I/DD), including people with Down syndrome.

The investigators are recruiting participants through collaboration with the New York State Office of People with Developmental Disabilities (OPWDD), Service Providers, Care Coordination Organizations and special programs, such as the Special Olympics. For participants who meet eligibility criteria and have consented or assented (as appropriate), a video call meeting is arranged to complete the baseline interview survey of socio-demographic characteristics and sexual and reproductive health knowledge and behaviors. The interview takes up to 45 minutes to complete. Once the baseline interview is completed the participant is randomly assigned to either the STEPS2 or the STYH arm of the study. Half of the participants will be randomized to STEPS2, and half to the STYH arm. Participants begin the intervention within 2 weeks of having completed the baseline survey.

For the intervention, participants in both arms receive virtual video call one hour weekly health education sessions for 6 weeks. The STEPS2 socialization and sexuality curriculum (experimental arm) is provided during one-on-one sessions between a Study Health Educator and the participant. The STYH curriculum (comparison arm) is provided during group sessions with 6-10 participants and a Study Health Educator. For both arms, participants choose whether they wish for a guardian or helper to also attend for a given session.

Participants have follow-up interview surveys at month 2 (after completing the health education intervention), month 6, and month 12, with the same sexual and reproductive health measures as included in the baseline survey. The month 2 interviews also include measures of participant satisfaction with the curriculum and with the Study Health Educator. Each survey takes up to 45 minutes to complete. Survey interviewers are blinded to which curriculum participants have received.

The investigators are comparing the proportion of participants who have had a conversation with a doctor about sex, know their HPV vaccination status, have had the HPV vaccine, and show an understanding of sex and pregnancy at the month 12 interview between the two arms, after adjusting for baseline measures of these indicators, to test whether participation in the STEPS2 arm had an effect on these measures. Analysis will include intention-to-treat estimates, as well as instrumental variable estimates to adjust for incomplete attendance to the 6-week curricula. Analyses will also be stratified by gender, age, and mild versus moderate I/DD.

If the STEPS2 curriculum is found to improve reproductive and sexual health knowledge and behaviors, the investigators will email the curriculum to all participants in the STYH arm at study completion. Both curricula will be made publicly available at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* 16-27 years of age
* resides in New York State
* mild/moderate I/DD
* willing to receive either STEPS2 or STYH curricula
* able to complete curriculum in English

Exclusion Criteria:

* if female sex, self-reports pregnant at screening

Ages: 16 Years to 27 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 856 (Estimated)
Dates: Start 2023-10-20 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Proportion who have had a sexual health discussion with medical professional | One year post enrollment
  Have had a sexual health discussion with medical professional
Proportion who know their HPV vaccination status | One year post enrollment
  Know whether they have been vaccinated for HPV
Proportion who have been vaccinated for HPV | One year post enrollment
  Have been vaccinated for HPV (self-report with verification using NYS and NYC immunization registry when possible)
Proportion who can accurately describe what sex is | One year post enrollment
  Understand what sex is based on response to an open-ended question
Proportion who can accurately describe how a person gets pregnant | One year post enrollment
  Can describe that vaginal sex can lead to pregnancy and the general mechanics of how this works in an open-ended question

SECONDARY OUTCOMES:
Average sexual health knowledge score (1-25, with 25 being high knowledge) | One year post enrollment
  Score based on sexual health knowledge survey questions
Average sexual health knowledge score (1-25, with 25 being high knowledge) | 6 months post enrollment
  Score based on sexual health knowledge survey questions
Average sexual health knowledge score (1-25, with 25 being high knowledge) | Two months post enrollment (after completion of 6 week intervention)
  Score based on sexual health knowledge survey questions
Proportion using birth control among those reporting vaginal sex | One year post enrollment
  Self-reported use of birth control among those reporting vaginal sex
Proportion using condoms among those reporting vaginal and/or anal sex | One year post enrollment
  Self-reported use of condoms among those reporting vaginal and/or anal sex
Proportion tested for STDs among those reporting vaginal and/or anal sex | One year post enrollment
  Self-reported STD testing among those reporting vaginal and/or anal sex
Average satisfaction with intervention score (1 to 5, with 5 being very satisfied) | Two months post enrollment (after completion of 6 week intervention)
  Average of self-reported satisfaction with 1. curriculum, 2. health educator and 3. participant manual (on a scale of 1 to 5 for each question)

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne McDermott, PhD, Principal Investigator — CUNY School of Public Health; Heidi E Jones, PhD, Principal Investigator — CUNY School of Public Health
Locations (1):
- CUNY School of Public Health (but interventions are virtual), New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Anonymized survey data from baseline, month 2, 6 and 12 will be made available for other researchers.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Anonymized data will be made available within 6 months of publication on primary endpoints, with no end date for this availability.
Access Criteria: We will make the data available on the NIH's Project INCLUDE data hub.
URL: https://portal.includedcc.org